CLINICAL TRIAL: NCT05494307
Title: A Multicenter Randomized Trial of Second Line Treatment for Corticosteroid-Resistant or Relapsed Immune Thrombocytopenia: Combined Terbutaline and Danazol Versus Danazol Monotherapy
Brief Title: The Combination of Terbutaline and Danazol as the Treatment of Corticosteroid-resistant/Relapse Immune Thrombocytopenia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice President of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PKU-ITP039
Record Dates: First submitted 2022-08-06; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Terbutaline; Danazol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terbutaline plus danazol (Experimental): Terbutaline: A dose of 2.5 mg three times daily for 16 weeks Danazol: A dose of 200 mg twice daily for 16 weeks
  Interventions: Drug: Terbutaline; Drug: Danazol
- Danazol monotherapy (Active Comparator): Danazol: A dose of 200 mg twice daily for 16 weeks
  Interventions: Drug: Danazol

INTERVENTIONS:
Drug: Terbutaline — Orally terbutaline at a dose of 2.5 mg three times daily for 16 weeks
  Arms: Terbutaline plus danazol
Drug: Danazol — Orally danazol at a dose of 200 mg twice daily for 16 weeks

SUMMARY:
A randomized, open-label, multicenter study to compare the efficacy and safety of terbutaline plus danazol compared to danazol monotherapy for the second-line treatment of adults with corticosteroid-resistant or relapsed primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicenter, randomized controlled trial of 228 adults with ITP in China. Patients were randomized to terbutaline plus danazol compared to danazol monotherapy group. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria: Patients >18 years old with corticosteroid-resistant or relapsed ITP who had either a platelet count of <30×10^9/L or a platelet count of <50×10^9/L and clinically significant bleeding.

1. Not achieving a sustained response to therapy with full-dose corticosteroids for a duration of at least 4 weeks or relapsed during the process of corticosteroid tapering or discontinuation;
2. Platelet counts <30×10^9/L or platelet counts < 50×10^9/L and significant bleeding symptoms (WHO bleeding scale 2 or above);
3. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Secondary ITP (have a known diagnosis of connective tissue diseases, malignancy, active infection, HIV infections or hepatitis B virus or hepatitis C virus infections);
3. Received drugs affecting the platelet counts within 6 months before the screening visit (e.g., chemotherapy, anticoagulants, etc);
4. Severe medical condition (lung, heart, hepatic or renal disorder);
5. Patients who are deemed unsuitable for the study by the investigator.
6. Patients who had hypertension, diabetes mellitus, hyperthyroidism or coronary heart disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall response | From date of randomization until 1 years or the end of follow-up
  Achieving a platelet count ≥ 30 × 10^9/L confirmed on at least two separate occasions (at least 7 days apart), at least a doubling of the baseline platelet count without any other ITP-specific treatment and the absence of bleeding.

SECONDARY OUTCOMES:
Sustained response | From date of randomization until 1 years or the end of follow-up
  maintenance of a platelet count > 30 × 10^9/L, an absence of bleeding, and no requirement for any other ITP-specific treatment for 6 consecutive months after achievement of OR
Complete response | From date of randomization until 1 years or the end of follow-up
  a platelet count ≥ 100 × 10^9/L measured on two occasions at least 7 days apart and the absence of bleeding
Remission | at 12-month follow-up
  a durable platelet count > 30 × 109/L without bleeding up to 12 months after randomization
Time to response | From date of randomization until 1 years or the end of follow-up
  the time from starting treatment to the time a response was achieved.
Duration of response | From date of randomization until 1 years or the end of follow-up
  time from OR until loss of response or until the last follow-up visit
Rescue therapy | From date of randomization until 1 years or the end of follow-up
  any new medical intervention taken to increase the platelet count or prevent bleeding events or an increase in the dose of concomitant treatments
Associated factors of treatment failure, OR, SR and remission | From date of randomization until 1 years or the end of follow-up
  Factors that are associated with treatment failure, OR, SR and remission
Number of patients with bleeding | From date of randomization until 1 years or the end of follow-up
  Number of patients with bleeding complication (WHO bleeding score)
Number of patients with side effects | From date of randomization until 1 years or the end of follow-up
  Number of patients with Medication adverse events.
Relapse | From date of randomization until 1 years or the end of follow-up
  Loss of OR
Relapse-free survival | From date of randomization until 1 years or the end of follow-up
  the time interval between achievement of OR and relapse or the end of the follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, MD, Principal Investigator — Peking University People's Hospital